CLINICAL TRIAL: NCT02043717
Title: Increasing Vitamin D Serum Levels Reduces Pulmonary Exacerbations in Patients With Cystic Fibrosis
Brief Title: Increased Vitamin D Reduces Pulmonary Exacerbations in CF
Status: Completed | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Other Study IDs: vitaminD-HMO-CTIL
Record Dates: First submitted 2014-01-12; First posted 2014-01-23 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Vitamin D; Lung function
MeSH Terms: conditions — Cystic Fibrosis | interventions — Vitamin D

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CF patients: Both children and adults, with or without vitamin D deficiency.
  Interventions: Dietary Supplement: Vitamin D

INTERVENTIONS:
Dietary Supplement: Vitamin D — Supplementing oral cholecalciferol according to the new guidelines by:
  Tangpricha V, Kelly a, Stephenson a, Maguiness K, Enders J, Robinson K a, et al. An update on the screening, diagnosis, management, and treatment of vitamin D deficiency in individuals with cystic fibrosis: evidence-based recommendations from the Cystic Fibrosis Foundation. The Journal of clinical endocrinology and metabolism [Internet]. 2012 May [cited 2012 Oct 31];97(4):1082-93. Available from: http://www.ncbi.nlm.nih.gov/pubmed/22399505

SUMMARY:
The investigators study is designed to test the hypothesis that correction of vitamin D in CF patients can increase their lung function and decrease the number of their pulmonary exacerbations.

DETAILED DESCRIPTION:
Vitamin D deficiency is a known problem in CF patients. The CF Foundation Committee published in April 2012 new guidelines for administering vitamin D in CF patients. The investigators' study is designed to look for association between normal serum vitamin D levels and lung function. ~100 CF patients from The Center of Chronic Diseases in Hadassah Medical Organization will be treated according to the new guidelines, and their lung function will be tested once a month during the trial, which will be held for at least one year. In this study, the investigators' goal is to test the efficiency of the new guidelines in correcting serum vitamin D levels, and to follow other related factors such as growth indices (height, weight, BMI), bone mineral density, number of pulmonary exacerbations and number of hospital admissions.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and laboratory diagnosis of Cystic Fibrosis
* Complete medical and nutritional follow-up for at least one year before changing the vitamin D dosage and follow up for at least one year afterwards.

Exclusion Criteria:

* Age under 4 years old (because of the inability to assess lung function in a reliable fashion)

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: CF patients (both children and adults) from The Center for Chronic Diseases in Hadassah Medical Organization.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
FEV1 (by % of predicted) | Baseline, and then, on average, once a month during trial (at least one year).
  Forced expiratory volume in the 1st second (by spirometry)

SECONDARY OUTCOMES:
Pulmonary Exacerbations (PEs) | Average number in a year
  Defined according to the research definition of the EuroCare CF Working Group - the need for additional antibiotic treatment as indicated by a recent change in at least two of the following: change in sputum volume, color or consistency, increased cough, increased malaise, fatigue or lethargy, increased dyspnea, anorexia or weight loss, decrease in FEV1 by ≥10% and/or presence of radiographic changes.
Days of Hospitalisation (DOHs) | Average number in a year
  Defined as days of admission to the hospital due to a CF-related complication such as pulmonary exacerbation, intravenous (IV) antibiotic treatment, pancreatitis, distal intestinal obstruction syndrome (DIOS), constipation and gastrointestinal bleeding or IV antibiotic treatment at home or as an outpatient at the CF Center.

OTHER OUTCOMES:
Vitamin D level | Baseline, and then, on average, once a month during trial (at least one year).
  Serum levels for 25(OH)D

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wilschanski, Prof., Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tangpricha V, Kelly A, Stephenson A, Maguiness K, Enders J, Robinson KA, Marshall BC, Borowitz D; Cystic Fibrosis Foundation Vitamin D Evidence-Based Review Committee. An update on the screening, diagnosis, management, and treatment of vitamin D deficiency in individuals with cystic fibrosis: evidence-based recommendations from the Cystic Fibrosis Foundation. J Clin Endocrinol Metab. 2012 Apr;97(4):1082-93. doi: 10.1210/jc.2011-3050. Epub 2012 Mar 7. PMID 22399505
- [Background] Green D, Carson K, Leonard A, Davis JE, Rosenstein B, Zeitlin P, Mogayzel P Jr. Current treatment recommendations for correcting vitamin D deficiency in pediatric patients with cystic fibrosis are inadequate. J Pediatr. 2008 Oct;153(4):554-9. doi: 10.1016/j.jpeds.2008.04.058. Epub 2008 Jun 27. PMID 18589445
- [Derived] Abu-Fraiha Y, Elyashar-Earon H, Shoseyov D, Cohen-Cymberknoh M, Armoni S, Kerem E, Wilschanski M. Increasing Vitamin D Serum Levels Is Associated With Reduced Pulmonary Exacerbations in Patients With Cystic Fibrosis. J Pediatr Gastroenterol Nutr. 2019 Jan;68(1):110-115. doi: 10.1097/MPG.0000000000002126. PMID 30095576